CLINICAL TRIAL: NCT03204955
Title: Low-chloride Versus High-chloride Containing Hypertonic Solution for the Treatment of Subarachnoid Hemorrhage-Related Complications
Brief Title: A Low ChloridE hyperTonic Solution for Brain Edema
Acronym: ACETATE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Owen Samuels, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00090456
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Subarachnoid Hemorrhage; Acute Kidney Injury
Keywords: Osmolar therapy; Acetate
MeSH Terms: conditions — Subarachnoid Hemorrhage; Acute Kidney Injury | interventions — Sodium Chloride; Sodium Acetate; Plasmalyte A

STUDY DESIGN:
Intervention Model Description: Once consented to the study, patients' serum chloride will be followed daily. Patients who will have a chloride concentration of 109mg/dL or above will be randomized to receive the blinded hypertonic solutions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blinded-double-dummy design, where each dose of hypertonic solution will be administered along with a balanced solution in order to mask the difference in the volume between the two solutions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium chloride /sodium acetate (16.4%) (Experimental): 50cc doses of sodium-chloride/sodium-acetate (16.4%) along with 30cc bag of dummy solution (PlasmaLyte).
  Interventions: Drug: Sodium chloride /sodium acetate (16.4%); Drug: PlasmaLyte
- Sodium chloride (23.4%) (Active Comparator): 30cc per dose of sodium chloride (23.4%) along with 50cc dummy solution bag (PlasmaLyte)
  Interventions: Drug: Sodium chloride (23.4%); Drug: PlasmaLyte

INTERVENTIONS:
Drug: Sodium chloride /sodium acetate (16.4%) — Sodium Acetate is a sterile, nonpyrogenic solution of Sodium Acetate intended as an alternative to sodium chloride to provide sodium ion in parenteral (IV) fluid therapy.
  Sodium Chloride is sterile, nonpyrogenic hypertonic saline (concentrated sodium-chloride) solution for parenteral (IV) fluid therapy.
  Arms: Sodium chloride /sodium acetate (16.4%)
Drug: Sodium chloride (23.4%) — Sodium Chloride is sterile, nonpyrogenic hypertonic saline (concentrated sodium-chloride) solution for parenteral (IV) fluid therapy.
  Arms: Sodium chloride (23.4%)
Drug: PlasmaLyte — PlasmaLyte is an isotonic IV solution that mimics human physiological plasma electrolyte concentrations, osmolality and pH.
  Other Names: Placebo solution

SUMMARY:
This pilot study will compare the two hypertonic solutions currently used for subarachnoid hemorrhage (SAH) - related complications and to determine if the reduction of chloride load is safer, and as efficacious as the classic hypertonic solution.

DETAILED DESCRIPTION:
This pilot study aimed to collect high-quality randomized and prospective information to help plan a future, larger multicenter trial. The study will compare the two hypertonic solutions currently used for subarachnoid hemorrhage (SAH) - related complications and to determine if the reduction of chloride load by using a sodium acetate and sodium chloride mixture can lead to a relative reduction of serum chloride, reduce kidney injury, and as efficacious as the classic hypertonic solution.

Hyperosmolar therapy is one of the mainstay treatments for SAH-related cerebral edema and vasospasm, in order to reduce delayed cerebral ischemia. Recent evidence from the literature correlates high chloride load when applying IV fluids with worse outcome in a variety of critically-ill patients. Hypertonic saline, with which most hyperosmolar treatment is done, contains a supra-physiologic chloride load. It is possible that by changing the hypertonic solution to a "chloride-lean" one, the study team would be able to reduce the side effects of hypertonic sodium-chloride without losing its efficacy in treating SAH-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous SAH with an identified aneurysmal source as identified on neuroimaging obtained at admission to Emory University Hospital or with imaging at an outside hospital
* Age ≥ 18 years

Exclusion Criteria:

* SAH related to non-aneurysmal vascular anomaly
* SAH thought due to trauma
* SAH occurring in relation to another medical procedure (cardiac catheterization, LVAD placement, etc.)
* SAH with a negative workup for cause ("angio-negative")
* Patients who arrive in a brain-death state or in a devastating clinical status that will be presumed to lead to brain death or early withdrawal of treatment
* Patient who suffer from end-stage renal disease at baseline and who are routinely treated with dialysis
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Difference between serum chloride level on randomization day and the peak afterwards | Baseline, up to once daily during a patient's stay in the ICU, and up to 90 days
  Serum chloride levels will be measured as part of standard of care. Difference between serum chloride level on randomization day and the peak afterwards will be calculated.

SECONDARY OUTCOMES:
Number of patients with acute kidney injury (AKI) | Patients' stay in the ICU, and up to 90 days
  AKI diagnosis will be done on the basis of clinical parameters (serum creatinine ≥ 1.5 times baseline or ≥0.3 mg/dl and urine output (<0.5 ml/kg/h for 6 hours) according to Kidney Disease Improving Global Outcomes (KDIGO). Number of patients with acute kidney injury (AKI) will be recorded.
All causes of in-hospital mortality. | Patients' stay in the ICU, and up to 90 days
  All causes of in-hospital mortality, including withdrawal of treatment or discharge to a hospice facility, will be recorded.
All causes of 90 day mortality. | Up to 90 days
  All causes of mortality, 90 days post admission day, including withdrawal of treatment or discharge to a hospice facility, will be recorded.
Change in intracerebral pressure (ICP) measured by ICP monitor following hypertonic treatment. | Continuous measurement as long as the patient has an indication for an ICP monitor, and up to 90 days
  Change in intracerebral pressure (ICP) following the administration of the hypertonic solution will be recorded.
Change in serum sodium level following the administration of the hypertonic solution. | Baseline, and daily during a patient's stay in the ICU, and up to 90 days
  Serum sodium levels will be measured as part of standard of care. Difference between serum sodium level on randomization day and the peak afterwards will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Owen Samuels, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital's Neurointensive Care Unit, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sadan O, Singbartl K, Kraft J, Plancher JM, Greven ACM, Kandiah P, Pimentel C, Hall CL, Papangelou A, Asbury WH, Hanfelt JJ, Samuels O. Low-chloride- versus high-chloride-containing hypertonic solution for the treatment of subarachnoid hemorrhage-related complications: The ACETatE (A low ChloriE hyperTonic solution for brain Edema) randomized trial. J Intensive Care. 2020 May 4;8:32. doi: 10.1186/s40560-020-00449-0. eCollection 2020. PMID 32391156
- [Derived] Sadan O, Samuels O, Asbury WH, Hanfelt JJ, Singbartl K. Low-chloride versus high-chloride hypertonic solution for the treatment of subarachnoid hemorrhage-related complications (The ACETatE trial): study protocol for a pilot randomized controlled trial. Trials. 2018 Nov 14;19(1):628. doi: 10.1186/s13063-018-3007-7. PMID 30428930